CLINICAL TRIAL: NCT05849623
Title: Optimal Resection Technique for Medium-sized (10-20mm) Colorectal Polyps: A Randomized Clinical Trial
Brief Title: Optimal Resection Technique for Medium-sized (10-20mm) Colorectal Polyps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Samir Grover, Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-041
Record Dates: First submitted 2023-04-03; First posted 2023-05-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: 10-20mm Colorectal Polyp
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endoscopic Mucosal Resection (EMR) (Active Comparator): Patients will have an electrosurgical grounding pad attached, and an Erbe VIO electrosurgical unit will be adjusted to the endoscopist's preferred EndoCut Q and Coagulation settings. The polyp will be injected submucosally with a saline and methylene blue solution, with or without epinephrine at endoscopist's discretion. Using a 15mm snare connected to the electrosurgical unit, the resection will be performed, with the initial cut including a margin of normal mucosa and subsequent cuts to ensure no residual polyp tissue remains. In case of intraprocedural bleeding, snare tip soft coagulation (STSC) or coagulation forceps may be used. The resection site will be examined and any remaining polypoid tissue will be resected. Endoclips may be used to close the defect if there is significant intraprocedural bleeding. The polyp will be retrieved (en bloc or piecemeal) using suction into a trap or RothNet.
  Interventions: Procedure: Endoscopic Mucosal Resection (EMR)
- Cold Endoscopic Mucosal Resection (C-EMR) (Active Comparator): The polyp will be positioned at the 6 o'clock position and injected submucosally with saline and methylene blue, with or without epinephrine. The size of the ensnared polyp will be limited to 10-15mm to make sure that the snare will cut through the tissue. If the snare encounters difficulty in cutting through, it will be loosened to release deeper tissue before being closed again. The base and margins of the resected polyp will be inspected for residual polyp, which will be resected using the same technique if found. The polyp will be retrieved (en bloc or piecemeal) using suction into a trap or RothNet.
  Interventions: Procedure: Cold Endoscopic Mucosal Resection (C-EMR)
- Underwater Endoscopic Mucosal Resection (U-EMR) (Active Comparator): In the Underwater EMR arm, the patient will be connected to an electrosurgical grounding pad, and an Erbe VIO electrosurgical unit with EndoCut Q and Coagulation settings will be adjusted to the endoscopist's preference. Water, instead of carbon dioxide, will be used to fill the colon. Submucosal injection will not be performed.The patient will be positioned for optimal polyp exposure, and a 15mm snare will be used. The snare will be opened and positioned with a margin of normal mucosa and used to cut the polyp, en bloc if possible. Piecemeal resection should ensure no residual polyp tissue remains. Snare tip soft coagulation or coagulation forceps may be used for intraprocedural bleeding. The base and margins of the resected polyp will be inspected for residual polyp and resected if necessary. Closure of the defect with endoclips may be considered if there is significant bleeding. The polyp will be retrieved (en bloc or piecemeal) using suction into a trap or RothNet.
  Interventions: Procedure: Underwater Endoscopic Mucosal Resection (U-EMR)

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection (EMR) — EMR will be used to resect an eligible medium-sized polyp found in patients from this arm.
  Arms: Endoscopic Mucosal Resection (EMR)
Procedure: Cold Endoscopic Mucosal Resection (C-EMR) — C-EMR will be used to resect an eligible medium-sized polyp found in patients from this arm.
  Arms: Cold Endoscopic Mucosal Resection (C-EMR)
Procedure: Underwater Endoscopic Mucosal Resection (U-EMR) — U-EMR will be used to resect an eligible medium-sized polyp found in patients from this arm.
  Arms: Underwater Endoscopic Mucosal Resection (U-EMR)

SUMMARY:
This study will investigate which resection technique (Endoscopic Mucosal Resection (EMR), cold EMR, or underwater EMR) leads to lower recurrence rates and less adverse events in patients with colorectal polyps (10-20mm).

DETAILED DESCRIPTION:
Endoscopic resection of colorectal polyps has previously been demonstrated to lower the incidence of colorectal cancer, a major cause of cancer-related mortality globally. By disrupting the progression of adenomas into carcinomas, polypectomy is essential in effectively lowering colorectal cancer mortality. There is currently a surplus of high-quality research on the best ways to remove large polyps (>20mm). For colorectal polyps of 10 to 20 mm, however, the best endoscopic resection method is unknown. Due to the lack of a standard polypectomy technique for the complete removal of medium-sized colorectal polyps, clinicians use a variety of methods according to their preferences and local resources. The historic gold standard of treatment for resecting polyps greater than 10 mm is hot endoscopic mucosal resection (EMR). The term "hot" refers to the use of electrocautery to cut through dense mucosal tissue, ablate remaining marginal dysplastic tissue, and prevent rapid bleeding through thermal vascular coagulation. However, adverse events such as perforation, prolonged bleeding, and post-polypectomy syndrome are all linked to electrocautery-induced damage. In contrast, cold snare polypectomy (CSP) and cold electrocautery minimal resection with injection (C-EMR-I) are alternative well-established techniques for the removal of polyps smaller than 10 mm, demonstrated to be associated with less delayed adverse effects than EMR. Underwater EMR (U-EMR), a novel technique developed in the last decade wherein water is instilled into the colon, allowing for submucosal fat to rise, elevating the lesion, and allowing mucosal resection in the absence of submucosal injectate. U-EMR may achieving higher en bloc resection rates, R0 resection rates, and lower recurrence rates. There are no specific recommendations for EMR of medium-sized polyps from gastroenterological and endoscopic societies globally.

The aim of this randomized control study is to compare the polyp recurrence rates and adverse events between cold snare EMR (C-EMR), hot EMR (H-EMR) and underwater EMR (U-EMR) for colorectal polyps in the size of 10-20mm.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or a legally authorized representative) provides informed consent
2. 18 years of age or older
3. Completion of the endoscopist-recommended bowel preparation
4. Presence of one eligible medium-sized polyp:

   * 10-20 mm in size
   * Paris classification of 0-IIa (flat, elevated lesion) on standard white light colonoscopy
   * JNET Type 1 or 2A on magnifying Narrow Band Imaging (NBI) suspecting a sessile serrated lesion, adenoma, or adenoma with low-grade dysplasia.

Exclusion Criteria:

1. Patient < 18 years old
2. Inability to provide informed consent
3. Inflammatory Bowel Disease,
4. Familial Polyposis
5. Pregnancy
6. Incomplete bowel preparation
7. Patients with ineligible lesion:

   * Paris classification of 0-Ip or 0-Is on standard white light colonoscopy,
   * JNET Type 1 suspecting a hyperplastic polyp, or Type 2B or 3 suspecting a high- grade dysplasia or adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Polyp Recurrence Rate | Polyp recurrence rate will be determined during the follow-up procedure performed 6-12 months after the initial colonoscopy.
  The primary outcome of this study is the polyp recurrence rate at follow-up between the three techniques. Recurrence is evaluated 6 to 12 months after initial colonoscopy with endoscopic evaluation and biopsy of the scar. If adenoma is suspected under high-definition white light and/or electronic/conventional chromoendoscopy, the operator will remove it by snare or bioptic forceps. Final histology will be used to define recurrence rate.

SECONDARY OUTCOMES:
Adverse Events | AEs will be evaluated in both the initial and follow-up procedures. The follow-up procedure will be performed 6-12 months after the initial colonoscopy. Relevant AEs that occur during the procedure and within one day post-procedure will be recorded.
  The secondary outcomes include the number of adverse events and time spent performing the resection technique. Adverse events are defined according to the ASGE lexicon for endoscopic AEs. Major adverse events, such as bleeding and perforation will be evaluated. Procedure-related bleeding is defined as hematochezia and/or melena requiring follow-up endoscopy for hemostasis or transfusion. Perforation is endoscopically diagnosed as a visible hole in the colon wall during the procedure or the presence of free air on abdominal imaging after the resection. The ASGE lexicon will be used for detailed definition and timing of AEs.
Procedural time | Completion times will be recorded at the time of procedure for both initial and follow-up colonoscopies (performed 6-12 months after the initial procedure). The time to complete the resection technique will be recorded during the first colonoscopy.
  Amount of time it takes to complete the colonoscopy (cecal intubation time and withdrawal time), and the amount of time taken to perform the resection technique. U-EMR start when the perimeter of the lesion is identified, and the device is fully inserted. C-EMR and EMR start at the time of injection. All techniques are considered finished when all lesion pieces are retrieved.

CONTACTS AND LOCATIONS:
Overall Officials: Kareem Khalaf, HBSc, MD, Study Director — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No